CLINICAL TRIAL: NCT00107705
Title: A Single-blind Phase I Study to Assess the Residual Allergenicity of Tree (Birch, Hazel and Alder) Pollen Allergoid Using Skin Prick Testing
Brief Title: Assessment of Residual Allergenicity of Tree (Birch, Hazel, and Alder) Pollen Allergoid Using Skin Prick Testing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TreeMATAMPL101; P1DP05001
Record Dates: First submitted 2005-04-07; First posted 2005-04-08 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Type I Hypersensitivity
Keywords: allergy; skin prick test; allergoid; allergenicity; specific immunotherapy
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

INTERVENTIONS:
Biological: Tree MATA MPL

SUMMARY:
The purpose of this study is to evaluate the residual allergenicity of Tree MATA (modified pollen allergen tyrosine adsorbate) by skin prick testing. This is done by a comparison of the wheal response after skin prick testing with aqueous native and modified allergen, modified tyrosine adsorbed allergen and Tree MATA MPL (modified tyrosine adsorbed + MPL [Monophosphoryl Lipid A]).

DETAILED DESCRIPTION:
Tree MATA MPL has been developed to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to cross reacting tree pollens. MPL (Monophosphoryl Lipid A), a purified, detoxified glycolipid derived from the cell wall of Salmonella minnesota, is included in the product formulation as an adjuvant to increase the immunogenic effect of the product and to enhance the switch from an allergen-specific TH2 to a TH1-like profile.

The tree pollen extract is modified with glutaraldehyde to produce the active ingredient, an allergoid. This modification reduces the reactivity of the extract with IgE antibody, thus reducing the risk of side effects. However, a simultaneous reduction in other important immunological properties, such as IgG and T cell reactivities is not seen.

The purpose of this study is to assess residual allergenicity of the modified tree pollen in Tree MATA MPL using skin prick testing.

ELIGIBILITY:
Inclusion Criteria:

* The subject must sign the study consent form prior to any screening procedures being performed.
* If the volunteer is female of childbearing potential, she must demonstrate a negative urine pregnancy test and agree to remain abstinent or use an effective method of birth control or use a hormonal contraceptive
* The subject must demonstrate a positive skin prick test to Birch, Hazel and Alder pollen allergen extract
* The subject must demonstrate a positive skin prick test to positive histamine control
* The subject must demonstrate a negative skin prick test to negative control
* The subject must demonstrate a specific IgE for Birch, Hazel and Alder as documented by a RAST (radioallergosorbent test), or equivalent test
* The subject must have clinically acceptable results from the screening procedure.

Exclusion Criteria:

* History or presence of acute or subacute atopic dermatitis, chronic dermatitis, urticaria factitia, or urticaria due to physical/chemical influence or any other skin conditions which might interfere with the interpretation of skin prick test results
* Visual inspection of the forearms indicates potential problems with the conduct or interpretation of the skin prick tests; both forearms must be available for testing
* Subject has asthma or other lower respiratory tract condition
* History or presence of diabetes, cancer or any clinically significant cardiac, metabolic, renal, hepatic, gastrointestinal, dermatologic, venereal, hematologic, neurologic or psychiatric diseases or disorders
* Any clinically significant abnormal laboratory value at Visit 1
* Clinically relevant sensitivity to any common perennial allergen: house dust mites, molds, epithelia (cat, dog, and horse), grass mix
* Clinically relevant symptoms due to an IgE - mediated allergy at screening and before inclusion to the treatment period.
* Secondary alteration at the affected organ.
* History of auto-immune diseases or rheumatoid diseases
* Subject has a medical condition that prohibits the use of adrenalin
* Subject has disorder of tyrosine metabolism
* Subject with diseases interfering with the immune response and have received medication, which could influence the results of this study
* Subject has acute or chronic infection
* History of anaphylaxis
* History of angioedema
* Subjects determined by the Investigator to have any medical condition that could jeopardize their health or prejudice the results
* History of hypersensitivity to the excipients of the study medication
* History of immunotherapy with tree allergen extracts
* Current therapy with ß-blockers
* Currently receiving anti-allergy medication or other drugs with antihistaminic activity
* Subject has a positive drugs of abuse screen at Visit 1
* Subject participated in a clinical trial with an investigational drug within the last 30 days
* Subject cannot communicate reliably with the Investigator or is deemed uncooperative or noncompliant
* Females who are pregnant, breastfeeding, or refuse to use a reliable method of birth control
* Subject received treatment with a preparation containing MPL during the past 12 months
* Use of prohibited medications or inadequate washout periods prior to screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2005-04; Study Completion 2005-05

PRIMARY OUTCOMES:
to assess the allergenicity of the modified tree (birch, alder, hazel) pollen allergoid using skin prick testing

SECONDARY OUTCOMES:
evaluation for potential late phase reactions; adverse events; clinical labs; vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Karl Jürgen Fischer von Weikersthal-Drachenberg, MD, Study Chair — Allergy Therapeutics
Locations (1):
- Allied Research International Inc., Mississauga, Ontario, Canada